CLINICAL TRIAL: NCT02531295
Title: Immunologic Response to Euphorbia Kansui Extract Powder Prepared as Tea in HIV-infected Antiretroviral Therapy (ART)-Suppressed Individuals: a Dose Escalation Study
Brief Title: Immunologic Response to Kansui in Treated HIV+ Individuals: a Dose Escalation Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pause on clinical trial enrollment due to grant funding cuts after COVID-19
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Utah (Other); amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Principal Investigator, Sulggi A. Lee, MD, PhD, Principal Investigator, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: University of Utah #00100155
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: HIV; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Kansui 1g per day x 1 day (Experimental): Study participants will be given 1 g of Euphorbia kansui extract powder prepared as tea for a total of 1 daily dose.
  Interventions: Drug: Euphorbia kansui extract powder prepared as tea
- Kansui 1g per day x 2 days (Experimental): Study participants will be given 1 g of Euphorbia kansui extract powder prepared as tea for a total of 2 consecutive daily doses.
  Interventions: Drug: Euphorbia kansui extract powder prepared as tea
- Kansui 1g per day x 3 days (Experimental): Study participants will be given 1 g of Euphorbia kansui extract powder prepared as tea for a total of 3 consecutive daily doses.
  Interventions: Drug: Euphorbia kansui extract powder prepared as tea

INTERVENTIONS:
Drug: Euphorbia kansui extract powder prepared as tea — 1 g of Euphorbia kansui extract powder, measured and reconstituted in 4 fluid ounces of boiled water allowed to cool and administered as tea, taken by mouth daily
  Other Names: Kansui

SUMMARY:
The purpose of this study is to determine the safety and bioactivity of an herbal supplement called "kansui," which contains several active ingredients such as ingenols that may have a role in helping clear HIV from the body. Kansui has been used in traditional Chinese medicine for centuries to treat various ailments such as for eliminating excess fluid in the abdomen or lungs, loosening phlegm from the chest, and relieving constipation. Based on preliminary in vitro data from our group, kansui extract powder is a potent activator of HIV transpcription in latently infected Jurkat cells. The investigators' hypothesis is that kansui extract powder prepared as tea will be safe and well-tolerated, elicit an in vivo immunologic response, and at the doses administered, increase HIV transcription in latently-infected cells among HIV-infected patients on suppressive antiretroviral therapy.

DETAILED DESCRIPTION:
Millions HIV-infected individuals are now receiving life-saving antiretroviral therapy (ART). However, mortality remains high, particularly in resource-limited countries. Chronic HIV-infected individuals demonstrate evidence of persistent immune activation despite ART, which is an independent predictor of mortality in this setting. Given the current absence of an effective HIV vaccine, finding a cure for HIV will have a large impact on the long-term health of treated HIV-infected individuals. The key challenge of HIV eradication strategies is the persistence of a small pool of resting memory CD4+ T cells that harbor latent replication-competent HIV, untouched by current ART. One potential strategy to eliminate this reservoir in a "shock and kill" approach in which latency reactivating agents (LRAs) are used to "shock" the virus out of these cells in order for the host immune response, ART, and/or additional immunomodulatory agents to then kill the virus-expressing cells. The goal of the current study is to evaluate the safety and in vivo biological response to an herbal supplement used in traditional Chinese medicine ("kansui)" that has potent in vitro latency reactivating capabilities. Kansui is an inexpensive, readily available herbal supplement prescribed for thousands of years in traditional Chinese medicine and contains active compounds such as ingenols that have been shown to reverse latency in an animal model. A semi-synthetic form of ingenol has been shown to potently reactivate latent simian immunodeficiency virus (SIV) in rhesus macaques and is currently undergoing early drug development. Though kansui has been studied extensively in traditional Chinese medicine, this herbal supplement has never been evaluated for biologic activity in HIV disease using Western scientific research methods. This pilot clinical trial will generate preliminary results regarding the safety and in vivo biologic activity of kansui. Promising results from this study may allow future larger studies which can evaluate the efficacy of this non-pharmacologic agent in the treatment of HIV disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV-1 infection in adults aged 18 years or older.
2. Continuous therapy with a DHHS recommended/alternative combination ART for least 36 months (at least 3 agents) at study entry with no regimen changes in the preceding 24 weeks.
3. Maintenance of undetectable plasma HIV-1 RNA (<40 copies/ml) for at least 36 months. Episodes of single HIV plasma RNA 50-500 copies.ml will not exclude participation if subsequent HIV plasma RNA is <40 copies/ml.
4. Two CD4+ T cell counts >350 cells/μl in the six months prior to screening.

Exclusion Criteria:

1. Pre-ART viral load <2000 copies/ml (HIV controllers)
2. Based on prior history and/or virologic testing, no alternative ART regimens are available in the event that the current ART regimen is compromised as a result of this study.
3. Recent hospitalization in the last 90 days.
4. Recent infection in the last 90 days requiring systemic antibiotics.
5. Recent vaccination within the last 8 weeks prior to study scree or any study blood draw.
6. Any known history of liver-related diseases including but not limited to: hepatic cirrhosis of decompensated chronic liver diseases; clinically active hepatitis B or C infection as evidenced by clinical jaundice or Grade 2 or higher liver function test abnormalities; any hepatic impairment, regardless of the graded liver function test abnormalities.
7. Any known history of gastrointestinal diseases including but not limited to: history of diarrheal illness requiring the use of anti-motility agents including inflammatory bowel disease, chronic diarrhea not otherwise specified; history of gastrointestinal bleeding with hemoglobin below 12.5 g/dL; history of gastric or duodenal ulcers; inflammatory gastrointestinal disease such as Crohn's disease or ulcerative colitis
8. Any renal disease (eGFR < 90 ml/min) or acute nephritis.
9. Screening hemoglobin below 12.5 g/dL.
10. Screening TSH consistent with hypothyroidism.
11. Significant myocardial disease (current myocarditis or reduced left ventricular ejection fraction below the lower limit of normal) or diagnosed coronary artery disease.
12. Significant respiratory disease requiring oxygen.
13. Diabetes or current hypothyroidism.
14. Participants of reproductive potential or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test at screening. All participants of childbearing potential must agree to use a double-barrier method of contraception throughout the study period and up to 90 days after the last dose of kansui.
15. Exposure to any immunomodulatory drug (including maraviroc) in the16 weeks prior to study.
16. Prior or current use of experiment agents used with the intent to perturb the HIV-1 viral reservoir.
17. History of seizures, psychosis, abnormal electroencephalogram or brain damage with significant persisting neurological deficit
18. Positive test for tuberculosis by either skin test (PPD) or blood interferon-gamma release assay (QuantiFERON).
19. Significant substance use, which in the opinion of the investigator(s), is likely to interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sulggi A Lee, MD PhD, Principal Investigator — University of California, San Francisco; Adam M Spivak, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Cary DC, Fujinaga K, Peterlin BM. Euphorbia Kansui Reactivates Latent HIV. PLoS One. 2016 Dec 15;11(12):e0168027. doi: 10.1371/journal.pone.0168027. eCollection 2016. PMID 27977742
- [Result] Wang P, Lu P, Qu X, Shen Y, Zeng H, Zhu X, Zhu Y, Li X, Wu H, Xu J, Lu H, Ma Z, Zhu H. Reactivation of HIV-1 from Latency by an Ingenol Derivative from Euphorbia Kansui. Sci Rep. 2017 Aug 25;7(1):9451. doi: 10.1038/s41598-017-07157-0. PMID 28842560
- [Result] Liu Q, Li W, Huang L, Asada Y, Morris-Natschke SL, Chen CH, Lee KH, Koike K. Identification, structural modification, and dichotomous effects on human immunodeficiency virus type 1 (HIV-1) replication of ingenane esters from Euphorbia kansui. Eur J Med Chem. 2018 Aug 5;156:618-627. doi: 10.1016/j.ejmech.2018.07.020. Epub 2018 Jul 19. PMID 30031972

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo 1g Per Day x 1 Day: Study participants will be given 1 g of placebo prepared as tea for a total of 1 daily dose.
- Placebo 1g Per Day x 2 Days: Study participants will be given 1 g placebo prepared as tea for a total of 2 consecutive daily doses.
- Placebo 1g Per Day x 3 Days: Study participants will be given 1 g of placebo prepared as tea for a total of 3 consecutive daily doses.
Period: Overall Study
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
Started | 2 | 0 | 1 | 0 | 0 | 2
Completed | 2 | 0 | 1 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — The study was terminated (Halted Prematurely). | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated (Halted Prematurely).
Groups:
- Total: Total of all reporting groups
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days | Total
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 |  |  | 0 | 0
  Between 18 and 65 years | 2 |  | 1 |  |  | 2 | 5
  >=65 years | 0 |  | 0 |  |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (6.4) |  | 56 (0) |  |  | 55.1 (4.4) | 49 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 0 |  |  | 1 | 2
  Male | 1 |  | 1 |  |  | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 |  |  | 0 | 0
  Asian | 0 |  | 0 |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 |  |  | 0 | 0
  Black or African American | 1 |  | 0 |  |  | 0 | 1
  White | 1 |  | 1 |  |  | 2 | 4
  More than one race | 0 |  | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 1 |  |  | 2 | 5
HIV VL<40 [Count of Participants; unit: Participants] | 2 |  | 1 |  |  | 2 | 5
CD4 T Cell Count [Mean (Standard Deviation); unit: cells/uL] | 914 (359.7) |  | 428 (0) |  |  | 745.5 (225.6) | 732.1 (333.1)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Euphorbia Kansui Extract Powder Prepared as Tea Assessed by the Number of Grade 2 or Higher Severity Adverse Events or Drug-related Laboratory Abnormalities That Exceed a Frequency of 5%
Description: The number of grade 2 or higher severity adverse events (AEs) or drug-related laboratory abnormalities that exceed a frequency of 5% over a 31 day study period.
Time Frame: 31 days
Population: The study was terminated (Halted Prematurely).
Measure: Count of Participants; unit: Participants
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Early T Cell Immune Activation (Change in Percent CD69+ CD4+ and CD8+ T Cells From Baseline to 9 Days)
Description: The change in early immune activation levels (as measured by the Change in Percent CD69+ CD4+ and CD8+ T cells) over a 9 day study period.
Time Frame: Baseline and 9 days
Population: The study was terminated (Halted Prematurely). We do not have data for the last participant in placebo 1g per day x 3 days group.
Measure: Mean (Standard Deviation); unit: percentage of T cells
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 1
percentage of T cells
  Change in Percent CD69+ CD4+ T Cells | -0.175 (0.445) |  | 0.5 (0) |  |  | 7.49 (0)
  Change in Percent CD69+ CD8+ T Cells | 0 (0.608) |  | -2.1 (0) |  |  | 5.7 (0)

3. Secondary Outcome: T Cell Immune Activation (Change in Percent CD38+HLA-DR+ CD4+ and CD8+ T Cells From Baseline to 9 Days)
Description: The change in immune activation levels (as measured by the percent change in CD38+HLADR+ CD4+ and CD8+ T cells) over a 9 day study period.
Time Frame: Baseline and 9 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of T cells
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 2
percentage of T cells
  Change in Percent CD38+HLA-DR+ CD4+ T Cells | 0.05 (0.03) |  | -0.11 (0) |  |  | 0.03 (0)
  Change in Percent CD38+HLA-DR+ CD8+ T Cells | 0.5 (0.72) |  | -0.3 (0) |  |  | 0.2 (0)

4. Secondary Outcome: HIV Reservoir Size (Change in HIV RNA Pol Levels in Copies/ug From Baseline to 9 Days)
Description: The change in HIV reservoir size (as measured by cell-associated unspliced ddPCR HIV RNA Pol levels in copies/ug) over a 9 day study period.
Time Frame: Baseline and 9 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: copies/ug
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 1
copies/ug | -0.17 (0.24) |  | -59.9 (0) |  |  | -10.9 (0)

5. Secondary Outcome: HIV Reservoir Size (Plasma HIV RNA Level From Baseline to 9 Days)
Description: The change in HIV reservoir size (as measured by ultra-sensitive plasma HIV RNA levels) over a 9 day study period.
Time Frame: Baseline and 9 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: copies/ug
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 1
copies/ug | -128.6 (139.44) |  | 56 (0) |  |  | -68.8 (0)

ADVERSE EVENTS:
Time Frame: The total duration of the study was approximately 10 months from May 15, 2019 to March 19, 2020. Each participant was assessed for 31 days during the duration of their enrollment in the study. No severe adverse events occurred during the trial. There were no discontinuations or participants who left the trial early.
Description: Systematic assessment through detailed questionnaires and principal investigator physical exam assessment was conducted at each visit.
Arm/Group | Kansui 1g Per Day x 1 Day | Kansui 1g Per Day x 2 Days | Kansui 1g Per Day x 3 Days | Placebo 1g Per Day x 1 Day | Placebo 1g Per Day x 2 Days | Placebo 1g Per Day x 3 Days
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/1 | 0/0 | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1 | 0/0 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1 | 0/0 | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT02531295/Prot_SAP_000.pdf